CLINICAL TRIAL: NCT06160453
Title: HEROES: Human Extremity Robotic Rehabilitation and Outcome Enhancement for Stroke
Acronym: HEROES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Professor, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 73297
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Chronic Stroke; Motor disability; Rehabilitation; Neuroplasticity; Robotics; Wearables
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study (Parallel Assignment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stroke with upper limb monoparesis or hemiparesis (Experimental): Patients from Greece, 18 y.o. or older, suffering from chronic stroke and motor disability
  Interventions: Device: Brain-Computer Interface control of robotic arms with augmented reality; Device: Serious game with augmented reality
- Stroke with monoplegia or hemiplegia (Experimental): Patients from Greece, 18 y.o. or older, suffering from chronic stroke and motor disability
  Interventions: Device: Brain-Computer Interface control of robotic arms with augmented reality; Device: Serious game with augmented reality
- Healthy Participants (Active Comparator): Healthy participants, age and sex matched to the participants in the other arms
  Interventions: Device: Brain-Computer Interface control of robotic arms with augmented reality; Device: Serious game with augmented reality

INTERVENTIONS:
Device: Brain-Computer Interface control of robotic arms with augmented reality — The participants will be trained to modulate self-paced Visual Motor Imagery (VMI) and Kinesthetic Motor Imagery (KMI) under EEG recording in order to achieve BCI-control of a custom-built bimanual arms robot (MERCURY v2.0). In KMI they will be asked to modulate brain waves in order to learn to control the BCI and in VMI they will additionally be projected a visual cue (representation of the intended movement). BCI will be used to control the arms in physical space as well as in an Augmented Reality Environment. Each participant will take part in 3 sessions
Device: Serious game with augmented reality — The participants will don wearable robotics and use them as input to play a dojo-themed immersive serious game intended at tracking participants movement and presenting them with motor tasks to perform. The game will be played in a computer screen, as well as in an Augmented Reality Environment. Each participant will take part in 10 sessions

SUMMARY:
HEROES is a multidisciplinary neurophysiological & neural rehabilitation engineering project, developed by the Lab of Medical Physics & Digital Innovation, School of Medicine, Faculty of Health Science Aristotle University of Thessaloniki and supported by a Neurosurgical Department. The website for the project can be accessed at https://heroes.med.auth.gr.

The investigation's primary objectives include the development, testing and optimization of an intervention based on multiple immersive man-machine interfaces offering rich feedback, that include a) mountable robotic arm controlled with wireless Brain-Computer Interface and b) wearable robotics jacket & gloves in combination with a serious game application and c) augmented reality module for the presentation of the previous two, as well as the development and validation of a self-paced neuro-rehabilitation protocol for patients after chronic stroke with severe residual motor disability.

DETAILED DESCRIPTION:
HEROES project's full title is <Human Extremity Robotic Rehabilitation and Outcome Enhancement for Stroke>. It is a multidisciplinary neurophysiological & neural rehabilitation engineering project, developed by the Lab of Medical Physics & Digital Innovation, School of Medicine, Faculty of Health Science Aristotle University of Thessaloniki and supported by a Neurosurgical Department. The website for the project can be accessed at https://heroes.med.auth.gr .

The HEROES project involves:

* A clinical study for rehabilitation of patients with Chronic Stroke (CS), using multiple immersive man-machine interfaces (Brain-Computer Interface (BCI) controlled robotic arms device, Wearable Robotics Jacket & Gloves, Serious Gaming Application, Augmented Reality presentation)
* A secondary off-line neurophysiological analysis of brain activation, connectivity and plasticity as well as muscle electrophysiology in patients with CS undergoing motor imagery (MI) and BCI training and assistance through electrical muscle stimulation

Milestones of the study:

* The investigators aim to develop, test and optimize an intervention based on multiple immersive man-machine interfaces
* The investigators aim to develop and validate self-paced neuro-rehabilitation protocols for patients with CS.
* The investigators aim to identify and study the neurophysiological functionality and alteration of brain activity in chronic CS.

The brain neuron networks of Chronic Stroke (CS) patients and healthy individuals share similar connectivity patterns of, but new functional interactions have been identified as unique to CS patient networks and can be attributed to both adaptive and maladaptive organization effects after the stroke. The importance of such phenomena both as possible prognostic factors and as contributors to patient rehabilitation remains unspecified yet. The exact underlying neurophysiological process and the extent that this is modulated by higher-order interactions is also not fully understood. The investigators used rich visual and tactile feedback, virtual reality environments (VRE), BCI controlled exoskeleton and robotic actuators and furthermore documented plasticity effects at the brain networks.

Retraining brain circuits and promoting plasticity to restore body functions have been recognized among key principles of spinal cord repair by the US National Institute of Neurological Disorders and Stroke (US NIH/NINDS). Nonetheless, existing literature does not yet portray with precision the pathophysiological process and effect of CS on Central Nervous System (CNS) and the sensorimotor networks. Studies needed to address this issue (such as our study) should be considered, identifying specific questions to be answered through further investigation: a) how and why reorganization of CNS networks is established, b) how this reorganization evolves in time with respect to the severity and chronicity of the stroke, c) when can it be considered an adaptive or maladaptive evolution, and d) how can it be promoted or prevented respectively. The gained insight is expected to hold clinical relevance in preventing maladaptive plasticity after CS through individualized neuro-rehabilitation, as well as in the design of assistive technologies for CS patients.

This HEROES study is a both a pre-clinical neurophysiological investigation on human CS patients that aims to advance basic knowledge on CS sequelae to CNS and also a translational implementation in clinical (rehabilitation) practice. Our analysis aims to eventually help produce a model of CNS function along different stages of stroke (Acute, Sub-acute, Chronic), during different activity (resting state, simple motor tasks, complex sensorimotor activity), and ideally being able to predict negative outcome versus possible Recovery. The HEROES project aims to investigate and promote dormant neuroplasticity after chronic stroke, a type of injury that causes hemiparesis, hemiplegia, tetraparesis or tetraplegia. Our protocol will deploy training in brain computer interfaces and robotic arms, virtual environments (brain-controlled virtual arms, avatars and augmented reality wearable robotics with sensors and actuators (gloves & jacket) and rich audio/visual/tactile stimuli along with serious gaming applications to enhance motivation. Visual and kinesthetic sensorimotor brain networks will also be studied using high density electroencephalography in order to demonstrate and monitor CNS plasticity.

This research project was supported by the Hellenic Foundation for Research and Innovation (H.F.R.I.) https://www.elidek.gr under the "2nd Call for H.F.R.I. Research Projects to support Faculty Members & Researchers" (Project number: 4391).

ELIGIBILITY:
Inclusion Criteria:

* At least 14 years of age
* Female & male stroke survivors and healthy individuals (age and gender matched)
* Sufficient documentation of stroke in case of patients (clinical neurological examination, MRI)

Exclusion Criteria:

* Other neurological condition that has a possibility to significantly affect the neurological status of the participants (or) the ability to control a BCI (or) the neurophysiological recordings:
* Traumatic brain injury
* Central Nervous System tumors
* Multiple Sclerosis
* Amyotrophic Lateral Sclerosis
* Parkinson's disease
* Refractory Epilepsy
* Other grave medical condition that could affect the participation (or) the safety of the participants:
* Cardiac deficiency
* Pulmonary deficiency
* Hearing and visual impairments that can affect the participant's understanding of the --intervention and performance.
* Illegal drug use
* Chronic alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
BCI control | 1 week
  The ability of participants to modulate brainwave activity in order to achieve control of the BCI will be established. BCI control is evaluated as achieved or not (there are cases of BCI-illiteracy when the participants cannot modulate their brainwaves in order to control the BCI).
Serious game performance (in-game scoring system) | 2 weeks
  The ability of participants to control the wearables robotic jacket in order to complete in-game tasks and collect more points will be evaluated. The points will be gathered be matching the speed and position of the in-game task instructions while receiving assistance from electrical muscle stimulation.

SECONDARY OUTCOMES:
Initial Functional Improvement (Greek translation of the Modified Rankin Scale (mRS-9Q) | 12 months
  Daily functionality as measured by the Greek translation of the Modified Rankin Scale (mRS-9Q). The scale ranges from 0 to 5, where 0 is the best.

CONTACTS AND LOCATIONS:
Overall Officials: Panos D Bamidis, PhD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Laboratory of Medical Physics and Digital Innovation, AUTH, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made available after a Memorandum of Understanding agreement between the Medical Physics and Digital Innovation lab of Aristotle University of Thessaloniki and any interested party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be made available 2 years after the conclusion of the study

REFERENCES:
- See also: Project webpage — https://heroes.med.auth.gr
- See also: Location webpage — https://imedphys.med.auth.gr